CLINICAL TRIAL: NCT06363422
Title: The Value of Epicanthoplasty on the Modification of Upper-eyelid Appearance: a Retrospective Study
Brief Title: The Value of Epicanthoplasty on the Modification of Upper-eyelid Appearance
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: JY2024-012
Record Dates: First submitted 2024-04-07; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Patient Satisfaction; Epicanthus; Fold
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical
  Interventions: Procedure: Epicanthoplasty

INTERVENTIONS:
Procedure: Epicanthoplasty — Patients with unsatisfied blepharoplasty underwent epicanthoplasty in our center

SUMMARY:
In East Asian populations, the combination of an epicanthic fold and mono-eyelid is one of their anatomical characteristics. Misalignment of the orbicularis oculi muscle and fibrous connections leads to longitudinal tension, forming the epicanthic fold. The epicanthic fold may diminish the aesthetic effects of eyelid cosmetic surgery, shorten the horizontal length, and affect the postoperative shape of double eyelids. As upper eyelid cosmetic surgery is one of the most common cosmetic procedures in Asia, there is increasing attention on the modification of the epicanthic fold and its impact on the formation of double eyelids.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients who have previously undergone unsatisfactory blepharoplasty, combined with epicanthic fold issues;

  2: Underwent epicanthoplasty in this center

  3: over 18-year-old and less than 60-year-old

  4: Clinical data was comprehensive.

Exclusion Criteria:

* 1: The patient has concurrent untreated lacrimal defects, excessive eyelid skin, and other complications such as entropion and ectropion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In East Asian populations, the combination of an epicanthic fold and mono-eyelid is one of their anatomical characteristic. The epicanthic fold may diminish the aesthetic effects of eyelid cosmetic surgery, shorten the horizontal length, and affect the postoperative shape of double eyelids
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
inter-epicanthal distance (IED) | preoperatively and through study completion, an average of 1 year
  The inter epicanthal distance was measured by the distance from left to right epicanthus.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, PhD., Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No